CLINICAL TRIAL: NCT06488599
Title: Marginal Bone Loss Around Mandibular Implant-retaining Overdentures and Implant Supported Fixed Hybrid Prosthesis: A 5-year Follow-up
Brief Title: Marginal Bone Loss Around Mandibular Implant-retaining Overdentures and Implant Supported Fixed Hybrid Prosthesis
Status: Enrolling by invitation | Type: Observational
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Other Study IDs: USJ-2023-20
Record Dates: First submitted 2024-06-24; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Bone Loss in Jaw; Dental Implant Failure Nos; Dental Implant Failed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1- hybrid prosthesis: Patients having fixed hybrid prosthesis over 4 implants in the mandible for 5 years
  Interventions: Radiation: Peri-apical radiographs on the implants
- 2- over denture: Patients having removable overdenture with locators over 2 implants in the mandible for 5 years
  Interventions: Radiation: Peri-apical radiographs on the implants

INTERVENTIONS:
Radiation: Peri-apical radiographs on the implants — Peri-apical radiographs on the implants supporting the prosthesis

SUMMARY:
Few if any studies have compared marginal bone loss (MBL) around implant-retaining overdentures (2 implants with locators) versus implant supported fixed hybrid prosthesis (over 4 implants) in the mandible.

DETAILED DESCRIPTION:
Material and Methods: Patients of the saint Joseph university dental clinics, who have already in their records peri-apical radiographs of the implants post loading, will be divided in 2 groups depending on the prosthetic treatment that they have had for 5 years in mouth, and will be recalled for a check-up session during which the investigators will take new peri-apical X-rays by means of the parallel long-cone technique for the implants that are supporting/retaining the prosthesis. A total of minimum 50 implants placed in a minimum of 19 patients will be examined. The mean mesial and distal radiographic MBL and bone to implant contact (BIC) will be recorded by comparing the two X-rays for each implant.

the investigators will also investigate the possibly related factors that may have contributed to this marginal bone loss such as the medical history, smoking habits, oral hygiene, compliance, presence of keratinized tissue and possibility of proper cleaning.

Results: the investigators aim to find a statistically significant difference in the Marginal bone loss around implants assisting these two types of prosthesis and a possible correlation with some risk and modifying factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with mandibular implant-retaining overdentures (2 implants)
* Patients treated with mandibular implant-supported fixed hybrid prosthesis (4 implants)
* Patients having in their records a post-loading peri-apical radiograph for the implants
* Patients who have had their prosthesis for 5 years in mouth

Exclusion Criteria:

* Patients treated with mandibular implant-retaining overdentures with more or less than 2 implants
* Patients treated with mandibular implant-supported fixed hybrid prosthesis with more or less than 4 implants Patients treated with any other prosthetic option on implants Patients who don't have a post-loading peri-apical radiograph in their records

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: To determine the sample size, a power analysis was conducted for independent Student t test using G*Power and considering a power = 80%, alpha = 5%, and an effect size = 1.06. The minimum sample size required for this study is 50 implants in total: (25 per group)
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Loss in mm (MBL) | 5 years
  MBL in mm around implants in patients having a removable prosthesis over locators and in patients having a screw retained hybrid prosthesis

SECONDARY OUTCOMES:
smoking status | 5 years
  non smoker, smoker less than 10 cig/day, smoker more than 10 cig/day
compliance and attendance to recall sessions | 5 years
  patient attending the recall sessions or no
keratinized tissue hight | 5 years
  measured in mm with a periodontal probe
framework design | 5 years
  prosthetic framework fit/misfit
age | 5 years
  in years
health status | 5 years
  diabetes yes/no ; cardiovascular disease yes/no
sex | 5 years
  male female
plaque score | 5 years
  using the modified plaque index (0 absence,1 detectable by a probe, 2 visible, 3 abundant)

CONTACTS AND LOCATIONS:
Overall Officials: Elies El Hachem, DDS, Principal Investigator — Saint Joseph University of Beirut, Faculty of dental Medicine, Periodontolgy department; Nadim Mokbel, PhD, Study Director — Saint Joseph University of Beirut, Faculty of dental Medicine, Periodontolgy department
Locations (1):
- Saint Joseph University of beirut, Beirut, Lebanon